CLINICAL TRIAL: NCT00954694
Title: Assessing the Impact of an Introductory Exercise Regimen: An Analysis of the Consequent Effects of NuStep in Relation to Physical Activity and Lifestyle Adjustment in Adults With Type 1 and Type 2 Diabetes
Brief Title: Analysis of the NuStep as an Introductory Fitness Regimen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nebraska (Other)
Responsible Party: Kristina Volkmer/exercise physiologist, The Nebraska Medical Center Diabetes Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 328-09-FB
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes; Inactivity
MeSH Terms: conditions — Diabetes Mellitus; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- introductory exercise regimen (Experimental): sedentary adults will be introduced to an introductory fitness regimen using the NuStep
  Interventions: Device: NuStep fitness apparatus

INTERVENTIONS:
Device: NuStep fitness apparatus — The NuStep is a mode of exercise that has recently been used in clinical settings to determine appropriate intensity recommendations and energy expenditures. The NuStep exercise implement provides simultaneous upper and lower body movement while in a seated position. The machine stimulates all major muscle groups while putting minimal strain on joints. Ten resistance settings are offered and the device is fully adjustable to accommodate users of varying sizes (NuStep, 2009).

SUMMARY:
The purpose of this research study is to determine if participation in a fifteen week introductory exercise regimen using the NuStep by sedentary adults diagnosed with Type 1 or Type 2 diabetes will affect exercise adherence and lifestyle adjustment. This study will examine if using the NuStep encourages participants to seek other modes and facilitates interest in exercise. Age, gender, weight, height, waist-to-hip ratio, heart rate, blood pressure, 6-minute walk test, and A1C will be recorded pre, mid-point, and post-test. During each NuStep exercise session heart rate, blood pressure, blood glucose level, oxygen saturation, METs, and the Borg rate of perceived exertion will be monitored.

Associations between NuStep use and exercise adherence are investigated through the following hypothesis and null hypothesis. There is an association between using the NuStep as an introductory exercise regimen by sedentary adults diagnosed with Type 1 or Type 2 diabetes and exercise adherence. The null hypothesis states there is no association between using the NuStep as an introductory exercise regimen by sedentary adults diagnosed with Type 1 or Type 2 diabetes and exercise adherence. The primary endpoint of the study is the qualitative measurement, by use of a questionnaire, of attitude and interest toward exercise in participants by assessing if they choose to seek and perform other modes of exercise. Secondary endpoints are the quantitative measurement of the change in weight, waist-to-hip ratio, heart rate, blood pressure, 6-minute walk test, and A1C levels.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults diagnosed by a physician with Type 1 diabetes or Type 2 diabetes. Sedentary adults are defined as persons 19 years of age and older that are not meeting the minimal physical activity recommendations from the U.S. Surgeon General's report.

Exclusion Criteria:

* Adults with:

  * severe cardiovascular disease (high blood pressure, abnormal heart rhythm, peripheral artery disease, atherosclerosis, congestive heart failure, congenital heart disease, valvular heart disease and coronary artery disease)
  * amputees
  * severe foot ulcers
  * severe neuropathy
  * an amplified susceptibility to hypoglycemia
  * those weighing 400 lbs. or more, or inability to adequately perform exercise

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the qualitative measurement, by use of a questionnaire, of attitude and interest toward exercise in participants by assessing if they choose to seek and perform other modes of exercise. | 15 weeks

SECONDARY OUTCOMES:
Secondary endpoints are the quantitative measurement of the change in weight, waist-to-hip ratio, heart rate, blood pressure, 6-minute walk test, and A1C levels. | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Volkmer, MPH, Principal Investigator — The Nebraska Medical Center
Locations (1):
- The Nebraska Medical Center Diabetes Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] American Diabetes Assocation. (2002). Handbook of exercise in diabetes. Alexandria, Virginia: Transcontinental Publishing. Coquart, J.B., Lemaire, C., Dubart A.,E., Luttembacher, D.P., Douillard, C., & Garcin, M. (2008). Intermittent versus continuous exercise :Effects of perceptually lower exercise in obese women. Medicine Science Sports Exercise, 40(8);1546-53. Conn, V., Vanetine, J., & Cooper, H. (2002). Interventions to Increase Physical Activity Among Aging Adults: A Meta-Analysis. The Annuals Of Behavioral Medicine, 24(3);190-200. Donahue, M.D. (2003). Physiological responses to submaximal workload on four exercise ergometers. Kinesiology Abstracts, 16(1). Glaros, N.M., & Janeele, C.M. (2001). Varying the mode of cardiovascular exercise to increase adherence. Journal of Sport Behavior, 24(2), 42-63. Gutbrod, N., Hiniker, J., Oakes, A., & Smecko, J. (2008). Physiological responses of the NuStep for individuals with cardiovascular disease. Journal of Undergraduate Kinesiology, Vol 3(2), 60-67. McCutcheon, S. (2008), Recumbent stepper: Aerobic testing and training protocol development. Masters Abstracts International. 45(6), 2008-2009. NuStep. (2009). Retrieved May 1, 2009, from http:///www.nustep.com/product/trs4000 Patten, C., Armstrong, C., Martin, J., Sallis, J., & Booth, J. (2000). Behavioral control of exercise in adults: Studies 7 and 8. Psychology and Health, 15, 571-581. Tantiwong, P., & Musi, N. (2009) The importance of exercise. Practical diabetology, 28(2). U.S. Department of Health and Human Services Office of the Surgeon General. (2009). Retrieved April 30, 2009 from http://www.health.gov/paguidelines/guidelines/summary.aspx Wasserman, K., Hansen, J.E., & Sue, D.Y., Principles of Exercise Testing. Philadelphia : Lea & Febiger, 1987 :79.